CLINICAL TRIAL: NCT00085553
Title: Phase I Trial of R115777 and OSI-774 in Patients With Advanced Solid Tumors
Brief Title: Tipifarnib and Erlotinib Hydrochloride in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02597; NCI-2012-02597 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000370818; NCI-6014; MAYO-MC0212; MC0212; MC0212 (Other: Mayo Clinic); 6014 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Solid Neoplasm
MeSH Terms: interventions — Erlotinib Hydrochloride; tipifarnib

ARMS (1):
- Treatment (erlotinib hydrochloride, tipifarnib) (Experimental): Patients receive erlotinib hydrochloride PO QD on days 1-28 (days 8-28 of course 1 as of 11/4/2013) and tipifarnib PO BID on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. (Closed to accrual as of 2/2/06)
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Tipifarnib

INTERVENTIONS:
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Tipifarnib — Given PO
  Other Names: R115777; Zarnestra

SUMMARY:
This phase I trial studies the side effects and best dose of tipifarnib and erlotinib hydrochloride in treating patients with solid tumors that have spread to other places in the body. Tipifarnib and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximal tolerated dose of R115777 (tipifarnib) in combination with OSI-774 (erlotinib hydrochloride).

II. To describe the toxicity profile of this combination. III. To evaluate the effect of OSI-774 on the disposition of R115777. IV. To evaluate in vitro markers of farnesyl transferase (FT) inhibition and epidermal growth factor receptor (EGFR) inhibition.

OUTLINE: This is a dose-escalation study.

Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-28 (days 8-28 of course 1 as of 11/4/2013) and tipifarnib PO twice daily (BID) on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. (Closed to accrual as of 2/2/06)

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is unresectable and for which no standard life-prolonging therapy is available
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet count (PLT) >= 100,000/uL
* Total bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Creatinine =< 1.5 x ULN
* Hemoglobin (Hgb) >= 9.0 g/dL
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester for follow up
* Life expectancy >= 12 weeks
* At maximum tolerated dose (MTD) only: tumor that is amenable for serial biopsy
* Medically capable and willing to provide the biologic specimens as required by the protocol Note: The goals of this study include assessment of the biologic effects on surrogate markers of the agent(s) being tested and are, therefore, contingent upon availability of the biologic specimens; patients with pre-existing clinical contraindications (e.g. anticoagulant therapy) for biopsy will be excluded from participation in the study; however, those patients who develop a major complication associated with the first biopsy (e.g. bleeding) or who develop clinical contraindications (e.g., anticoagulant therapy) after entry on study may remain on the study without the requirement for further tissue biopsies; this stipulation only applies to the 12 patients enrolled in Cohort II at MTD; the stipulation for provision of biologic specimens, as noted above, excludes the optional pharmacogenomic specimen

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 2, 3, or 4
* Uncontrolled infection
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks prior to study entry
  * Mitomycin C/nitrosoureas =< 6 weeks prior to study entry
  * Immunotherapy =< 4 weeks prior to study entry
  * Biologic therapy =< 4 weeks prior to study entry
  * Hormonal cancer therapy =< 4 weeks prior to study entry
  * Radiation therapy =< 4 weeks prior to study entry
  * Radiation to > 25% of bone marrow
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Patients on enzyme-inducing anticonvulsants (Phenobarbital, Dilantin, or Tegretol)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (condoms plus spermicidal agents, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.)
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Prior treatment with EGFR targeting therapies (e.g., ZD-1869, EKB-569, OSI-774, CI-1033, GW572016, C225, EMD72000) or Farnesyl transferase inhibitors (R115777, SCH66336, BMS2146632)
* Major surgery, or significant traumatic injury occurring =< 21 days prior to study entry
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjögren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Gastrointestinal tract disease resulting in an inability to take oral or nasogastric medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy
* Known brain metastases unless treated with surgery and/or radiation and stable for >= 8 weeks; patient should not be on enzyme-inducing anticonvulsants (Phenobarbital, Phenytoin (Dilantin) or Carbamazepine (Tegretol))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-05-20 (Actual); Primary Completion 2008-05-07 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Incidence of all adverse events, graded according to the National Cancer Institute Common (NCI) Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 30 days after last study treatment
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Incidence of toxicity graded according to NCI CTCAE version 3.0 | Up to 3 months
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.

SECONDARY OUTCOMES:
Best response as assessed by the Response Evaluation Criteria in Solid Tumors | Start of the treatment until disease progression/recurrence, assessed up to 3 months
  Best Response is defined to be the best objective status recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Time until any treatment related toxicity | Up to 30 days after last study treatment
Time until treatment related grade 3+ toxicity | Up to 30 days after last study treatment
Time until hematologic nadirs (white blood cells, ANC, platelets) | Up to 3 months
Time to progression | Up to 3 months
Time to treatment failure | Time from registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months

OTHER OUTCOMES:
Inhibition of EGFR from tumor biopsies | Up to day 21 of course 1
  Any change in these measures will be summarized descriptively within each patient and as whole group.
Inhibition of FT from tumor biopsies | Up to day 21 of course 1
  Any change in these measures will be summarized descriptively within each patient and as whole group.
Incidence of any genetic polymorphisms | Up to day 21 of course 1
  Assessed and summarized descriptively in those patients treated at the MTD.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Molina, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States